CLINICAL TRIAL: NCT01713608
Title: A Randomised, Placebo-controlled, Dose-escalation Study to Investigate Safety and Toleration of OZ439 OD for 3 Days to Healthy Male and Female Volunteers
Brief Title: A Dose-escalation Study to Investigate Safety and Toleration of OZ439
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Medicines for Malaria Venture (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: MMV_OZ439_12_005; 2012-004187-22 (EudraCT Number)
Record Dates: First submitted 2012-10-22; First posted 2012-10-25 (Estimated); Results first posted 2015-03-23 (Estimated); Last update posted 2015-03-23 (Estimated); Status verified 2015-03

CONDITIONS: Malaria
Keywords: malaria; dose escalation; safety; tolerability; maximum tolerated dose
MeSH Terms: conditions — Malaria

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- OZ439 Dose level 1 (300mg) (Experimental): • Cohort 1 (12 subjects: 8 Active [A] and 4 on Placebo [P]) Active dose will consist of 300mg OZ439 drinking solution administered once daily for 3 days
  Interventions: Drug: OZ439
- OZ439 Dose level 2 (Experimental): • Cohort 2 (12 subjects: 8 A, 4P). Subjects on active will receive X amount of OZ439 (dose level to be determined based on safety and tolerability of previous dose level) drinking solution once daily for 3 days
  Interventions: Drug: OZ439
- OZ439 dose level 3 (Experimental): Cohort 3 (12 subjects: 8 A, 4P). Subjects on active will receive X amount of OZ439 (dose level to be determined based on safety and tolerability of previous dose level) drinking solution once daily for 3 days
  Interventions: Drug: OZ439

INTERVENTIONS:
Drug: OZ439 — OZ439 x mg once daily for 3 days with milk

SUMMARY:
A randomised, placebo-controlled, dose-escalation study to investigate safety and toleration of OZ439 OD for 3 days to healthy male and female volunteers. The study aims:

* To determine the safety and tolerability of ascending doses of OZ439 OD for three days.
* To assess pharmacokinetic parameters of ascending doses of OZ439 given OD.
* To identify the maximum tolerated dose of OZ439 administered.

DETAILED DESCRIPTION:
This study will be conducted in a randomised, placebo-controlled dose-escalation design with OZ439 OD administered with full fat milk for three days to healthy male and female subjects between 18 to 55 years of age, using features of an adaptive study design. The study is expected to have three cohorts with a total of 36 healthy male and female subjects. An additional two cohorts may be used if required. The results of this study will inform the maximum tolerated exposure of OZ439 following OD dosing for three days in subjects who are not fasted.

ELIGIBILITY:
Inclusions:

1. healthy males or females of any race aged 18 - 55 years
2. BMI of 18 - 30 kg/m2 inclusive at screening
3. Agree to use acceptable methods of contraception if of childbearing potential
4. Capable of understanding and complying with the requirements of the protocol and must have signed the informed consent form
5. Females are either of child bearing potential or are confirmed as post-menopausal. Post-menopausal is defined as being amenorrheic for 12 months without an alternative medical cause with a screening FSH level ≥ 25.8 IU/L

Exclusions:

1. Male subjects with female partner(s) who is (are) pregnant or lactating from the time of the first administration of study medication
2. Clinically significant disease or any condition or disease that might affect drug absorption, distribution or excretion
3. History of allergic reactions to artemisinin-based compounds or any other clinically relevant allergy to drugs or food
4. Clinically relevant history of both soya and cow's milk intolerance/allergy
5. Clinically significant abnormal laboratory, vital signs or other safety findings as determined by medical history, physical examination or other evaluations conducted at screening or on admission
6. Electrocardiogram (ECG) abnormalities in the standard 12-lead ECG (at screening) and/or 24-hour 5 lead Holter ECG (at screening)
7. Any abnormalities in rhythm, conduction or morphology of resting ECG that may interfere with the interpretation of QTc interval changes
8. Prolonged QTcF >450 ms or shortened QTcF <340 ms, or family history of Long QT Syndrome
9. History or current evidence of any clinically relevant cardiovascular, pulmonary, hepatic, renal, gastrointestinal, haematological, endocrinological, metabolic, neurological, psychiatric, or other disease
10. Positive results in any of the serology tests for Hepatitis B Surface Antigen (HbsAg), anti Hepatitis core antibody (anti HBc Ig G [and anti HBc IgM if IgG is positive], Hepatitis C antibodies (anti HCV), and HIV 1 and 2 antibodies (anti HIV 1/2)
11. Confirmed positive results from urine drug screen (amphetamines, benzodiazepines, cocaine, cannabinoids, opiates, barbiturates, and methadone) or from the alcohol breath test at screening and on admission
12. History or clinical evidence of alcohol or drug abuse. Alcohol abuse is defined as regular weekly intake of more than 21 units for males and 14 units for females; drug abuse is defined as compulsive, repetitive and/or chronic use of drugs or other substances with or without problems related to their use and/or where stopping or a reduction in dose will lead to withdrawal symptoms
13. Is pregnant or lactating (female subjects who are of childbearing potential must have negative pregnancy tests at screening and admission)
14. Mentally handicapped
15. Participation in a drug trial within 90 days prior to first drug administration
16. Use of any medication (incl. over-the-counter (OTC) medication) within 2 weeks prior to drug administration (Day 1) or within less than 10 times the elimination half-life of the respective drug, or anticipated concomitant medication during the treatment periods, (whichever is longer), including herbal, traditional and alternative medications. Excluding oral contraceptives (combination oestrogen/progesterone pills), injectable progesterone or subdermal implants. Limited amounts (4g/day for 2 days) of paracetamol will be permitted for the treatment of AEs
17. Treatment with herbal supplements during the 7 days prior to drug administration, or use of vitamins during 48 hours prior to drug administration
18. Is not permitted to use strong inhibitors and/or inducers of CYP450 within 21 days prior to the planned first drug administration
19. Subjects have veins unsuitable for intravenous puncture or cannulation on either arm (e.g. veins that are difficult to locate, access or puncture veins with a tendency to rupture during or after puncture)
20. Blood ALT, AST and bilirubin should be in the normal range at screening and on admission
21. Donation of more than 500 mL of blood within 90 days prior to drug administration
22. Subjects must be non-smokers for at least three months prior to first drug administration
23. Any circumstances or conditions, which, in the opinion of the PI, may affect full participation in the trial or compliance with the protocol
24. Legal incapacity or limited legal capacity at screening
25. Subjects who are vegetarians, vegans or have any dietary restrictions conflicting with the study standardised menus

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 34 (Actual)
Dates: Start 2012-11; Primary Completion 2013-02 (Actual); Study Completion 2013-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Fiona Macintyre, PhD, Study Director — Medicines for Malaria Venture
Locations (1):
- Richmond Pharmacology Ltd, Croydon, Croydon, United Kingdom

RESULTS

PARTICIPANT FLOW:
Groups:
- OZ439 300mg: 300mg OZ439 drinking solution administered once daily for 3 days with milk
- OZ439 600mg: 600mg OZ439 drinking solution administered once daily for 3 days with milk
- OZ439 700mg: 700mg OZ439 drinking solution administered once daily for 3 days with milk
- Placebo: Placebo to match OZ439 PIB for oral suspension
Period: Overall Study
Arm/Group | OZ439 300mg | OZ439 600mg | OZ439 700mg | Placebo
Started | 8 | 6 | 8 | 12
Completed | 8 | 6 | 8 | 12
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: 34 subjects were enrolled with all 34 completing the study.
Groups:
- Total: Total of all reporting groups
Arm/Group | OZ439 300mg | OZ439 600mg | OZ439 700mg | Placebo | Total
Number analyzed (Participants) | 8 | 6 | 8 | 12 | 34
Age, Continuous [Mean (Standard Deviation); unit: years] | 30.5 (8.91) | 25.5 (3.39) | 33.4 (8.09) | 30.5 (7.24) | 30.3 (7.51)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 4 | 4 | 7 | 19
  Male | 4 | 2 | 4 | 5 | 15
Region of Enrollment [Number; unit: participants]
  United Kingdom | 8 | 6 | 8 | 12 | 34
Body Mass Index [Mean (Standard Deviation); unit: kg/m2] | 23.1 (2.99) | 22.4 (3.29) | 24.4 (2.78) | 24.2 (3.02) | 23.7 (2.97)

OUTCOME MEASURES:

1. Primary Outcome: OZ439 Cmax
Description: OZ439 maximum measured plasma concentration
Time Frame: Blood for analysis of OZ439 will be collected at the following times: pre-dose, 2, 4, 6, 8, 12, and 18 hours post-dose Day 1and Day 3, pre dose Day 2 and 4 hours post dose Day 2, and 24, 48, 72, 96 and 168 hours post 3rd dose and at follow up.
Population: PK Population: All subjects who received at least one dose of study medication and who had available evaluable PK data.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | OZ439 300mg | OZ439 600mg | OZ439 700mg
Number analyzed (Participants) | 8 | 6 | 8
ng/mL | 672 (183) | 1720 (544) | 1870 (600)

2. Secondary Outcome: OZ439 Tmax
Description: Time to reach maximum measured OZ439 plasma concentration
Time Frame: pre-dose, 2, 4, 6, 8, 12, and 18 hours post-dose Day 1and Day 3, pre dose Day 2 and 4 hours post dose Day 2, and 24, 48, 72, 96 and 168 hours post 3rd dose and at follow up.
Population: PK Population: All subjects who received at least one dose of study medication and who had available evaluable PK data.
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | OZ439 300mg | OZ439 600mg | OZ439 700mg
Number analyzed (Participants) | 8 | 6 | 8
hours | 3.26 (1.04) | 3.67 (0.816) | 4.00 (1.07)

3. Primary Outcome: OZ439 AUCτ
Description: OZ439 Area under the plasma concentration vs time curve from time zero to the time of the last quantifiable concentration t calculated using a log-linear trapezoidal method
Time Frame: as for outcome 2
Population: PK Population: All subjects who received at least one dose of study medication and who had available evaluable PK data.
Measure: Mean (Standard Deviation); unit: ng*h/mL
Arm/Group | OZ439 300mg | OZ439 600mg | OZ439 700mg
Number analyzed (Participants) | 8 | 6 | 8
ng*h/mL | 5970 (1340) | 16500 (5630) | 21300 (6250)

4. Secondary Outcome: OZ439 t½
Description: OZ439 estimated terminal phase half life
Time Frame: as for outcome 2
Population: PK Population: All subjects who received at least one dose of study medication and who had available evaluable PK data.
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | OZ439 300mg | OZ439 600mg | OZ439 700mg
Number analyzed (Participants) | 8 | 6 | 8
hours | 122 (36.2) | 130 (21.8) | 134 (44.5)

ADVERSE EVENTS:
Description: The safety analysis included all 34 subjects who had received at least one treatment of randomised study medication and for whom any post-treatment data was available.
Arm/Group | OZ439 300mg | OZ439 600mg | OZ439 700mg | Placebo
Serious Adverse Events (participants affected / at risk) | 0/8 | 0/6 | 0/8 | 0/12
Other Adverse Events (participants affected / at risk) | 3/8 | 2/6 | 6/8 | 5/12
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | OZ439 300mg (N=8) | OZ439 600mg (N=6) | OZ439 700mg (N=8) | Placebo (N=12)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Migraine (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Somnolence (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 0 (0) | 1 (1)
Upper respiratory tract infection (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 4 (4) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pregnancy (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Influenza like illness (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No